CLINICAL TRIAL: NCT06594029
Title: Community Participation Navigators: Testing a Peer Intervention for Adults With Serious Mental Illnesses
Brief Title: Community Navigators
Acronym: Navigators
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90IFRE0061; 31035 (Other: Temple University)
Record Dates: First submitted 2024-07-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Loneliness; Social Isolation; Mental Health Issue
Keywords: peer support; community participation; Serious Mental Illness
MeSH Terms: conditions — Social Isolation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Data analyst, research assistant conducting research interviews at baseline and post-treatment will be blind to participant allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Navigator Intervention (Experimental): Weekly meetings between participant and a peer specialist. The peer specialist will help participants identify participation interests, set participation goals, and to achieve those goals while increasing confidence and competence in community participation. Initially, participants will develop a plan for community participation which includes a list of meaningful activities, identifying potential barriers and facilitators to participation. At each weekly meeting, the peer specialist will work with participants to determine what aspects of the plan are working and modify it based on any newly identified barriers, opportunities, or changes to the participants' interests or motivation. The sessions are designed to meet the participants where they are on their journey towards participating in the community. Each successive session will encourage growth and independence through peer support that is tailored to each participant's particular needs and ability.
  Interventions: Behavioral: Community Navigator Intervention
- Active control group (Active Comparator): Receive information on community participation for adults with your health condition
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Community Navigator Intervention — see previous section
  Arms: Community Navigator Intervention
Other: Control Group — Participants receive information on how to increase their community participation
  Arms: Active control group

SUMMARY:
The Temple University Collaborative on Community Inclusion (TU Collaborative) is testing a community navigation intervention study based upon effective health navigation models by conducting a randomized controlled trial of the intervention to establish feasibility, efficacy, and outcomes among adults with serious mental illness (SMI).

DETAILED DESCRIPTION:
The study is a randomized, controlled trial (RCT) that will examine the effectiveness of an intervention designed to support and enhance community participation for adults with serious mental illness (SMI) receiving community mental health services. The intervention is based on two evidence-based strategies. The first is the patient navigation interventions, which are used to assist people with SMI to identify and overcome barriers to accessing care. The second is the Capability, Opportunity, Motivation model of behavior change (COM-B model) which evaluates how each of these factors influences behavior. Participants will be assigned to one of two groups, the Community Navigator condition, or a control group. Those in the intervention arm will develop a community support plan with a peer support specialist community navigator and those in the control arm will receive printed information on the importance, skills, and opportunities for participation. Over the course of the 6-month intervention, participants in the intervention arm, with support from the peer support specialist will develop an initial participation plan, and through weekly meetings online or in-person will monitor their progress and make changes as needed. Recruitment will occur only in Philadelphia in collaboration with residential treatment service providers including: Merakey, Horizon House, COMHAR, Inc, and potential others. Data collection for all participants will take occur at baseline and at the end of the 6-month intervention. We aim to recruit and enroll 96 participants for a 16-month period in a randomized control trial of a community navigation intervention. Participants will be randomly assigned to either the intervention or an informational control group. The intervention group will meet with a peer support specialist once a week for 60-90 minutes. Enrollment will occur over 16 months, with 6 participants joining each month from behavioral health residential service sites. Each participant will have two meetings with a research assistant - an intake interview and an exit interview after 6 months. The primary analyses are expected months after the study initiation.

The aim of the research study is to determine the efficacy of a peer-support intervention to navigate community opportunities and resource to increase participation among adults with SMI and to determine if participation in the intervention increases social connections and decreases loneliness. The existing navigation approaches in health care have employed peer-delivered services and demonstrated significant effects. The program theory of this intervention is based on existing models of peer-delivered health navigation approaches.

ELIGIBILITY:
Inclusion Criteria:

1. meet the criteria for an SMI diagnosis of schizophrenia, schizoaffective, bipolar, or major depression diagnosis based on the MINI,
2. are over the age of 18-years-old
3. are fluent in English: As current intervention materials and research and intervention personnel are only fluent in English, only participants who can communicate in written and spoken English are eligible for enrollment.
4. have a permanent residence without constraints on participation (free to come and go from residence without restrictions) 2
5. have the ability to provide informed consent.

Exclusion Criteria:

* inability to provide consent (legal guardian)
* unable to speak and understand English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Temple University Community Participation Scale (TUCP): | baseline, and post-treatment after 6 months
  self-reports of community participation in 22 different areas including going to a supermarket, participating in a community social group (like a book club or recreational sports team), going to a movie, or working for pay. Participants are asked to indicate the number of days in the past 30 days that they participated in each of the 22 areas, whether each participation area was important to them, and whether they felt they participated in each area enough, not enough, or too much. Recent research has found the measure to be reliable and valid. An updated version of this measure is included which adds questions related to relationships with intimate partners and children and digital participation.
WHO Disability Assessment Schedule | baseline, and post-treatment after 6 months
  measures each person's capability to participate. It assesses abilities in the areas of cognition, mobility, self-care, life activities, and participation. It contains 15-items.

SECONDARY OUTCOMES:
Clinical Assessment Interview for Negative Symptoms | baseline, and post-treatment after 6 months
  assesses motivation and pleasure. It is a 13-item interview that asks questions about motivation for relationships, school and work, and recreation activities. It also measures the frequency of pleasurable social activities, school and work activities, and recreation activities.
Assessment Opportunity | baseline, and post-treatment after 6 months
  will be done through a series of 12 questions that focus on both social and structural opportunities for participation. Social opportunities refer to having someone to go with and structural opportunities are related to environmental factors such as transportation, time, and resources.
The Social Embeddedness Scale | baseline, and post-treatment after 6 months
  subscale of the social network questionnaire (Shaw et al., 2007) that is used to identify degrees of social contact. It contains six items focused on social contact (e.g., visits, conversations) with friends and family in the previous two weeks.
Interpersonal Mattering Scale (Moschella & Baynard, 2021; Elliott et al., 2004): | baseline, and post-treatment after 6 months
  This 12-item scale examines three dimensions of mattering, including awareness ( α=.87), importance (α =.89), and reliance (α =.86).
3-Item UCLA Loneliness Scale (Hughes, Waite, Hawkley, & Cacioppo, 2004) | baseline, and post-treatment after 6 months
  This brief measure of loneliness has shown satisfactory reliability and validity in the measurement of overall loneliness.
Lehman Quality of Life Interview (QLI) | baseline, and post-treatment after 6 months
  assesses the overall quality of life of people with mental illness through an interview. There are 11 items that across three domains: community inclusion, holistic health and functioning, and human and legal rights. The statement "[If homeless or in jail, the place where you typically sleep at night?]" will be removed from Q5 the questionnaire as it is not relevant to our study participants.
Recovery Assessment Scale (RAS-20): | baseline, and post-treatment after 6 months
  assesses self-determination and hope as it relates to recovery. It is frequently used as an outcome measure for program evaluations. It is a 20-item self-report measure. Items are scored on a 5-point Likert scale and range from strongly agree to strongly disagree
The MOS Social Support survey | baseline, and post-treatment after 6 months
  A 19-item measure with 4 support scales (Emotional/Informational, Tangible, Affectionate, and Positive Social Interaction) and an overall functional social support index that has been shown to have good reliability and validity.

IPD SHARING:
Plan to Share IPD: Yes
All participants in the study will be required to complete informed consent forms which will include a clause about data preservation and sharing. Subjects will be assured that their identity will be protected and that no personally identifiable information (PII) will be disclosed as part of any data sharing.
  All data will be stored on Temple University's password protected, HIPAA-approved secure data server. However, because not all investigators who will need access to the data are at Temple, deidentified, anonymized data may be shared with other investigators via a secure file transfer system.
  All data in the study transferred between Temple University and collaborating institutions will be transferred through TUSafeSend using data encryption by way of a secure socket transfer protocol. TUSafeSend provides a secure method for transferring files containing confidential or other sensitive information, including HIPAA authorized data with PHI or PII.